CLINICAL TRIAL: NCT01100502
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of SGN-35 and Best Supportive Care (BSC) Versus Placebo and BSC in the Treatment of Patients at High Risk of Residual Hodgkin Lymphoma Following Autologous Stem Cell Transplant
Brief Title: A Phase 3 Study of Brentuximab Vedotin (SGN-35) in Patients at High Risk of Residual Hodgkin Lymphoma Following Stem Cell Transplant (The AETHERA Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGN35-005; 2009-016947-20 (EudraCT Number)
Expanded Access: NCT01196208 (No longer available)
Record Dates: First submitted 2010-04-06; First posted 2010-04-09 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Disease, Hodgkin
Keywords: Antigens, CD30; Antibody-Drug Conjugate; Antibodies, Monoclonal; Disease, Hodgkin; Drug Therapy; Hematologic Diseases; Immunotherapy; Lymphoma; Monomethylauristatin E
MeSH Terms: conditions — Hodgkin Disease; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brentuximab vedotin (Experimental): brentuximab vedotin 1.8 mg/kg every 3 weeks by IV infusion
  Interventions: Drug: brentuximab vedotin
- Placebo (Placebo Comparator): placebo every 3 weeks by IV infusion
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: brentuximab vedotin — Every 21 days by IV infusion (1.8 mg/kg)
  Other Names: SGN-35; Adcetris
  Arms: Brentuximab vedotin
Drug: placebo — Every 21 days by IV infusion
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter phase 3 trial to evaluate the efficacy and safety of brentuximab vedotin (SGN-35) and best supportive care (BSC) compared to placebo and BSC in treatment of residual Hodgkin lymphoma (HL) following autologous stem cell transplant (ASCT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with HL who have received ASCT in the previous 30-45 days
* Patients at high risk of residual HL post ASCT
* Histologically-confirmed HL
* ECOG of 0 or 1
* Adequate organ function

Exclusion Criteria:

* Previous treatment with brentuximab vedotin
* Previously received an allogeneic transplant
* Patients who were determined to have a best clinical response of progressive disease with salvage treatment immediately prior to ASCT
* History of another primary malignancy that has not been in remission for at least 3 years
* Post ASCT or current therapy with other systemic anti-neoplastic or investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2010-04-30 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2020-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lisano, PharmD, Study Director — Seagen Inc.
Locations (87):
- United States (32):
  - City of Hope National Medical Center, Duarte, California
  - University of California at San Francisco, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Section of Hematology/Oncology Lymphoma Program, Chicago, Illinois
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - Indiana University School of Medicine Simon Cancer Center 535 Barnhill Drive, RT 380, Indianapolis, Indiana
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York University Cancer Institute, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - UNC Lineberger Comprehensive Cancer Center / University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, The, Cleveland, Ohio
  - James Cancer Hospital / Ohio State University, Columbus, Ohio
  - Oregon Health and Science University / Center for Hematologic Malignancies, Portland, Oregon
  - Temple Bone Marrow Transplant Program, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Saint Francis Hospital, Greenville, South Carolina
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Bulgaria (2):
  - Specializirana bolnica aktivno lechenie detsa ohcohematologichni zabolyavania Hematologichno, Sofia
  - Specializirana bolnica za aktivno lechenie na hematologichni zabolyavania, Sofia
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove-oddeleni klinicke hematologie, Hradec Králové
  - Fakultni nemocnice Kralovske Vinohrady-oddeleni klinicke hematologie, Prague
  - Vseobecni fakultni nemocnice v Prahe-I. interni klinika, Prague
- France (5):
  - CHU Nantes - Hopital Hotel Dieu Service Hematologie, Nantes
  - Service des Maladies du Sang / Hospital Saint Louis, Paris
  - CHU Bordeaux Hopital Haut-Levaque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel / Centre Regional de Lutte Contre le Cancer, Rouen
- University Hospital of Cologne, Cologne, Germany
- Hungary (4):
  - Szent Istvan es Szent Laszlo Korhaz Rendelointezet Haematologiai es Ossejt-transzplantacios osztaly, Budapest
  - Debreceni Egyetem Orvos és Egeszsegtudomanyi Centrum, III. sz. Belgyogyaszati Klinika, Debrecen
  - Medical Center of the University of Pecs, 1st Clinic for Internal Medicine, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikat Kozpont, Szeged
- Italy (3):
  - Instituto di Ematologia ed Oncologia Medica, Bologna
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Istituto Nazionale dei Tumori, Milan
- Poland (9):
  - Klinika Hematologii i Transplantologii, Uniwersyteckie Centrum Kliniczne, Gdansk
  - Oddzial Transplantacji Szpiku Centrum Onkologii- Instytut M. Sklodowskiej-Curie, Oddzial Gliwicach, Gliwice
  - Samodzielny Publiczny Szpital Kliniczny im. Andrzeja Mieleckiego Slaskiego Uniwersytetu Medycznego, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Klinika Hematologii, Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi, Lodz
  - Oddzial Hematoonkologii, Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie, Lublin
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Klinika Hematologii, Instytut Hematologii i Transfuzjologii, Warsaw
  - Centrum Onkologii Institut im. Marii Sklodowskiej-Curie, Warsaw
- Romania (4):
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Sectia Clinica Hematologie si Transplant Medular, Târgu Mureş, Mureș County
  - Spitalul Clinic de Urgenta pentru Copii Louis Turcanu, Clinica III Pediatrie, Timișoara, Timiș County
  - Fundeni Clinical Institute, Bucharest
  - Institutul Clinic Fundeni, Centrul de Hematologie si Transplant Medular Stefan Berceanu, Bucharest
- Russia (12):
  - Burdenko Central Military Clinical Hospital, Moscow
  - Rossijskij onkologicheskij nauchnyj centr im. N.N. Blokhina RAMN, Moscow
  - Federal Medical Biophysical Center n.a. A.I. Burnazyan, Moscow
  - Gematologicheskj nauchnyj centr RAMN, Moscow
  - Uchrezhdenie Rossijskoj nauk Nauchno-issledovatel'skij institut klinicheskoj immunologii, Novosibirsk
  - Respublikanskaja bol'nica im. V.A. Baranova, Petrozavodsk
  - Leningradskaja oblastnaja klinicheskaja bol'nica, Saint Petersburg
  - Sankt-Peterburgskij gosudarstvennyj medicinskij universitet im. akademika I. P. Pavlova, Saint Petersburg
  - St. Petersburg Pavlov State Medical University, Saint Petersburg
  - Gorodskaya bol'nica #31, Saint Petersburg
  - Federal Center of Heart, Blood and Endocrinology n.a. V.A. Almazov under the Federal Agency for High, Saint Petersburg
  - Sverdlovskaja oblastnaja klinicheskaja bol'nica #1, Yekaterinburg
- Serbia (3):
  - Klinicki centar Srbije, Klinika za hematologiju, Belgrade
  - Vojnomedicinska akademija, Klinika za hematologiju, Belgrade
  - Klinicko bolnicki centar "Vojvodina", Klinika za hematologiju, Novi Sad
- Spain (5):
  - Complejo Hospitalano de Navarra Servicio Hematologia, Pamplona, Navarre
  - Hospital de la Santa Creu i Sant Paul, Barcelona
  - Hospital Clinic i Provincial Servicio Hematologia, Barcelona
  - Centro Oncologico MD Anderson, Madrid
  - Hospital Universitaro de Salamanca, Salamanca
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge
  - St James University Hospital, Leeds
  - Guy's Hospital Haematology Department, 4th Floor Southwark Wing, London
  - Christie Hospital NHS Foundation Trust, Manchester

REFERENCES:
- [Result] Moskowitz CH, Nademanee A, Masszi T, Agura E, Holowiecki J, Abidi MH, Chen AI, Stiff P, Gianni AM, Carella A, Osmanov D, Bachanova V, Sweetenham J, Sureda A, Huebner D, Sievers EL, Chi A, Larsen EK, Hunder NN, Walewski J; AETHERA Study Group. Brentuximab vedotin as consolidation therapy after autologous stem-cell transplantation in patients with Hodgkin's lymphoma at risk of relapse or progression (AETHERA): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2015 May 9;385(9980):1853-62. doi: 10.1016/S0140-6736(15)60165-9. Epub 2015 Mar 19. PMID 25796459
- [Derived] Moskowitz CH, Walewski J, Nademanee A, Masszi T, Agura E, Holowiecki J, Abidi MH, Chen AI, Stiff P, Viviani S, Bachanova V, Sureda A, McClendon T, Lee C, Lisano J, Sweetenham J. Five-year PFS from the AETHERA trial of brentuximab vedotin for Hodgkin lymphoma at high risk of progression or relapse. Blood. 2018 Dec 20;132(25):2639-2642. doi: 10.1182/blood-2018-07-861641. Epub 2018 Sep 28. PMID 30266774

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Apr 2010-Aug 2014
Period: Overall Study
Arm/Group | Brentuximab Vedotin | Placebo
Started | 165 | 164
Completed | 89 (Completed due to study closure by sponsor) | 70 (Completed due to study closure by sponsor)
Not Completed | 76 | 94
Not completed — Withdrawal by Subject | 18 | 25
Not completed — Lost to Follow-up | 13 | 28
Not completed — Site request to end participation in study | 0 | 1
Not completed — Death | 45 | 40

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Brentuximab Vedotin | Placebo | Total
Number analyzed (Participants) | 165 | 164 | 329
Age, Continuous [Median (Full Range); unit: years] | 33 [18 to 71] | 32 [18 to 76] | 32 [18 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 67 | 156
  Male | 76 | 97 | 173
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 2 | 12
  White | 153 | 156 | 309
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Russian Federation | 20 | 19 | 39
  Romania | 4 | 6 | 10
  Hungary | 9 | 11 | 20
  United States | 67 | 68 | 135
  United Kingdom | 3 | 3 | 6
  Spain | 4 | 6 | 10
  Czech Republic | 5 | 0 | 5
  Poland | 26 | 28 | 54
  Italy | 9 | 7 | 16
  France | 8 | 5 | 13
  Serbia | 3 | 6 | 9
  Bulgaria | 7 | 2 | 9
  Germany | 0 | 3 | 3
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead
  Participants
    0 | 87 | 97 | 184
    1 | 77 | 67 | 144
    2 | 1 | 0 | 1
Hodgkin Lymphoma Status after end of Frontline Therapy [Count of Participants; unit: Participants]
  Refractory | 99 | 97 | 196
  Relapse in less than 12 months | 53 | 54 | 107
  Relapse 12 months or later with extranodal disease | 13 | 13 | 26
Best Response to Salvage Therapy pre-ASCT [Count of Participants; unit: Participants]
  Complete remission | 61 | 62 | 123
  Partial remission | 57 | 56 | 113
  Stable disease | 47 | 46 | 93

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival by Independent Review
Description: Time from date of randomization to the first documentation of disease progression by independent review or to death due to any cause, whichever comes first
Time Frame: Up to approximately 4 years
Population: Intention-to-Treat analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin | Placebo
Number analyzed (Participants) | 165 | 164
months | 42.9 [30.4 to 42.9] | 24.1 [11.5 to NA] — Follow-up is not long enough to estimate an upper bound for median progression-free survival
Statistical Analysis 1: Comparison: Brentuximab Vedotin vs Placebo; Test type: Superiority or Other; p = 0.001, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.40 to 0.81]

2. Secondary Outcome: Overall Survival
Description: Time from date of randomization to date of death due to any cause
Time Frame: Up to approximately 10 years
Population: Intention-to-Treat analysis set
Measure: Median (Full Range); unit: months
Arm/Group | Brentuximab Vedotin | Placebo
Number analyzed (Participants) | 165 | 164
months | NA [1.31 to 117.88] — Due to patients lost to follow up, patient withdrawal of consent and post ASCT therapies; there were less deaths on study than anticipated. Therefore, median OS was not reached. | NA [0.03 to 119.23] — Due to patients lost to follow up, patient withdrawal of consent and post ASCT therapies; there were less deaths on study than anticipated. Therefore, median OS was not reached

3. Secondary Outcome: Incidence of Adverse Events or Laboratory Abnormalities
Time Frame: Up to 12 months
Population: Safety Analysis Set includes all patients who received at least 1 dose of brentuximab vedotin or only received placebo: 2 patients randomized to placebo received a single dose of brentuximab vedotin and are included in the brentuximab vedotin arm; 2 patients randomized to placebo received no study treatment and are not included in the analysis
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin | Placebo
Number analyzed (Participants) | 167 | 160
participants
  Any Treatment-Emergent Adverse Event | 163 | 142
  Any Treatment-Related Adverse Event | 147 | 79
  Any Adverse Event with Severity >= Grade 3 | 93 | 51
  Any Serious Adverse Event | 41 | 20
  Any Treatment-Related Serious Adverse Events | 19 | 7
  Treatment Discontinuation Due to Adverse Event | 54 | 10
  Any Laboratory Abnormalities Severity >=Grade 3 | 69 | 29

4. Secondary Outcome: Incidence of Anti-therapeutic Antibodies (ATA) to Brentuximab Vedotin
Time Frame: Up to 12 months
Population: ATA-evaluable patients (patients with a baseline and at least 1 postbaseline sample)
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin | Placebo
Number analyzed (Participants) | 157 | 154
participants
  Baseline Negative | 138 | 142
  Baseline Negative: -'ve Postbaseline | 92 | 104
  Baseline Negative: Transiently +'ve Postbaseline | 36 | 27
  Baseline Negative: Persistently +'ve Postbaseline | 10 | 11
  Baseline Positive | 19 | 12
  Baseline Positive: -'ve Postbaseline | 7 | 0
  Baseline Positive: Transiently +'ve Postbaseline | 9 | 5
  Baseline Positive: Persistently +'ve Postbaseline | 3 | 7

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were followed for up to 15 months. Serious adverse event data were collected for up to approximately 10 years (116 months).
Description: Safety Analysis Set includes all patients who received at least 1 dose of brentuximab vedotin or only received placebo: 2 patients randomized to placebo received a single dose of brentuximab vedotin and are included in the brentuximab vedotin arm; 2 patients randomized to placebo received no study treatment and are not included in the analysis
Arm/Group | Placebo | Brentuximab Vedotin
All-Cause Mortality (participants affected / at risk) | 40/160 | 45/167
Serious Adverse Events (participants affected / at risk) | 21/160 | 43/167
Other Adverse Events (participants affected / at risk) | 127/160 | 151/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=160) | Brentuximab Vedotin (N=167)
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 4
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 5
Asthenia (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 6
Hepatotoxicity (Hepatobiliary disorders) | 1 | 3
Acute hepatitis b (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Hepatic candidiasis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 2
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 7
Septic shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basilar migraine (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Radiation myelopathy (Injury, poisoning and procedural complications) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=160) | Brentuximab Vedotin (N=167)
Anaemia (Blood and lymphatic system disorders) | 4 | 14
Leukopenia (Blood and lymphatic system disorders) | 3 | 9
Neutropenia (Blood and lymphatic system disorders) | 18 | 58
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 12
Sinus tachycardia (Cardiac disorders) | 3 | 9
Abdominal pain (Gastrointestinal disorders) | 5 | 20
Constipation (Gastrointestinal disorders) | 5 | 20
Diarrhoea (Gastrointestinal disorders) | 15 | 33
Dyspepsia (Gastrointestinal disorders) | 6 | 11
Nausea (Gastrointestinal disorders) | 12 | 34
Vomiting (Gastrointestinal disorders) | 11 | 24
Asthenia (General disorders) | 7 | 13
Chills (General disorders) | 8 | 17
Fatigue (General disorders) | 29 | 40
Non-cardiac chest pain (General disorders) | 9 | 6
Oedema peripheral (General disorders) | 10 | 8
Pain (General disorders) | 5 | 11
Pyrexia (General disorders) | 23 | 27
Bronchitis (Infections and infestations) | 10 | 10
Herpes zoster (Infections and infestations) | 3 | 10
Pharyngitis (Infections and infestations) | 4 | 8
Sinusitis (Infections and infestations) | 10 | 4
Upper respiratory tract infection (Infections and infestations) | 37 | 43
Weight decreased (Investigations) | 9 | 31
Weight increased (Investigations) | 14 | 5
Decreased appetite (Metabolism and nutrition disorders) | 9 | 20
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 30
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 15
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 18
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 11
Headache (Nervous system disorders) | 13 | 18
Paraesthesia (Nervous system disorders) | 2 | 16
Peripheral motor neuropathy (Nervous system disorders) | 3 | 37
Peripheral sensory neuropathy (Nervous system disorders) | 25 | 92
Anxiety (Psychiatric disorders) | 13 | 14
Insomnia (Psychiatric disorders) | 5 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 21
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 10
Night sweats (Skin and subcutaneous tissue disorders) | 18 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 22
Rash (Skin and subcutaneous tissue disorders) | 5 | 14
Hypotension (Vascular disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less